CLINICAL TRIAL: NCT01243541
Title: Cold Therapy to Prevent Paclitaxel-Induced Peripheral Neuropathy and Cutaneous Toxicity
Brief Title: Cryotherapy in Preventing Peripheral Neuropathy and Nail Toxicity in Patients With Breast Cancer Who Are Receiving Paclitaxel
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decision due to low accrual and lack of funding
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NU 10CC03; NCI-2010-02105; STU00033028 (Other: Northwestern University IRB)
Record Dates: First submitted 2010-10-29; First posted 2010-11-18 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Chemotherapeutic Agent Toxicity; Pain; Peripheral Neuropathy; Recurrent Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer; Therapy-related Toxicity
MeSH Terms: conditions — Pain; Peripheral Nervous System Diseases; Breast Neoplasms | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients wear an Elasto-Gel cold glove and sock on their dominant hand and foot every two weeks on days the patient is scheduled for paclitaxel.The glove and sock is worn for 15 minutes prior to paclitaxel infusion, 3 hours during treatment, and for 15 minutes after completion of chemotherapy for a total of 210 minutes.
  Interventions: Procedure: cryotherapy; Other: questionnaire administration; Procedure: quality-of-life assessment; Procedure: management of therapy complications; Procedure: assessment of therapy complications
- Arm II (Experimental): Patients wear an Elasto-Gel cold glove and sock on their non-dominant hand and foot every two weeks on days the patient is scheduled for paclitaxel. The glove and sock is worn for 15 minutes prior to paclitaxel infusion, 3 hours during treatment, and for 15 minutes after completion of chemotherapy for a total of 210 minutes.
  Interventions: Procedure: cryotherapy; Other: questionnaire administration; Procedure: quality-of-life assessment; Procedure: management of therapy complications; Procedure: assessment of therapy complications

INTERVENTIONS:
Procedure: cryotherapy — Patients wear an Elasto-Gel cold glove and sock
Other: questionnaire administration — Ancillary studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Procedure: management of therapy complications — In this therapeutic study, cold therapy is administered with an Elasto-Gel cold glove and sock (study device) that will be worn on your right hand and foot or your left hand and foot. The study device is a glycerine-based gel cold pack shaped like a mitten or sock with a cloth-like fabric kept at a constant temperature. The study device is not known to cause any major adverse affects and it is considered of non-significant risk. If you choose to participate in this study, you will be asked to wear a glove and sock at each paclitaxel infusion (4 treatments total). We hope the use of this study device will prevent or significantly reduce the onset and potential severity of paclitaxel-induced peripheral neuropathy and nail problems.
  Other Names: complications of therapy, management of
Procedure: assessment of therapy complications — Study Treatment Assessment You will be asked permission for pictures to be taken of only your hands and feet. This is to have a visual documentation of symptom development during your treatment. This will be done at all six time points before you begin chemotherapy that day.

SUMMARY:
RATIONALE: Cryotherapy may help prevent peripheral neuropathy or nail toxicity in patients receiving chemotherapy. PURPOSE: This clinical trial studies cryotherapy in preventing peripheral neuropathy and nail toxicity in patients with breast cancer who are receiving paclitaxel.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. Differences in "tingling" and "numbness" (measured on 0-10 numeric rating scale; as measured by NPSI) between treated and untreated extremities at conclusion of paclitaxel therapy). SECONDARY OBJECTIVES: I. Differences in nail toxicity between treated and untreated extremities as measured by NCI-CTC v4.0 from baseline to conclusion of taxane therapy and at each time point (after each infusion and at conclusion of taxane therapy). II. Differences in peripheral sensory neuropathy subscale of NCI-CTC v 4.0 between treated and untreated extremities at each time point (after each infusion and at conclusion of paclitaxel therapy). III. Differences in pain intensity (0-10 from BPI) between treated and untreated extremities at each time point (after each infusion and at conclusion of paclitaxel therapy). IV. Differences in quantitative sensory testing between treated and untreated extremities at each time point (after each infusion and at conclusion of paclitaxel therapy). OUTLINE: Patients are randomized to 1of 2 treatment arms. ARM I. Patients wear an Elasto-Gel cold glove and sock on their dominant hand and foot every two weeks on days the patient is scheduled for paclitaxel.The glove and sock is worn for 15 minutes prior to paclitaxel infusion, 3 hours during treatment, and for 15 minutes after completion of chemotherapy for a total of 210 minutes. ARM II: Patients wear an Elasto-Gel cold glove and sock on their non-dominant hand and foot every two weeks on days the patient is scheduled for paclitaxel. The glove and sock is worn for 15 minutes prior to paclitaxel infusion, 3 hours during treatment, and for 15 minutes after completion of chemotherapy for a total of 210 minutes. In both arms, treatment repeats every 2 weeks for 4 courses in the absences of unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically confirmed diagnosis of breast cancer (any stage)
* Must be receiving either adjuvant or neo-adjuvant dose-dense anthracycline/taxane-based chemotherapy
* Specifically, this study seeks to characterize neuropathies associated with patients receiving paclitaxel cycles separated by two week intervals
* Patients may have received any of the following therapies: surgery, chemotherapy, hormones, biologics, or radiation
* Prior chemotherapies are permitted, except with prior treatments with taxanes
* Required lab values: CBC, Comprehensive Chemistry Panel
* Desired lab values: If the patient's record also includes TSH, HbA1c, and folate, then those will be recorded as well
* All patients will have given signed, informed consent prior to registration

Exclusion Criteria:

* Patients must not have received any prior taxane treatments
* Patients must not have a history of peripheral neuropathy (regardless of cause)
* Patient must not have a history of diabetes mellitus
* Patient must not have a history of Raynaud's disease
* Men are not eligible

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-11-03 (Actual); Primary Completion 2014-04-04 (Actual); Study Completion 2014-04-04 (Actual)

PRIMARY OUTCOMES:
To assess the primary aim of the study to determine the differences in "tingling" and "numbness" (measured on a 0-10 numeric rating scale) between the treated and untreated extremities. | Periodically during study treatment
To compare the treated or untreated extremities with respect to the percentage having score values of 4 or greater. | After completion of study treatment

SECONDARY OUTCOMES:
To compare the treated and untreated extremities at each time point with respect to the ratings in regards to the NCI-CTC v4.0, BPI, and QSTs. | Periodically during study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Judith Paice, PhD, RN, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States